## **INFORMED CONSENT FORM [Feasibility Trial- Stage 3]**

## Official title: Developing a self-persuasion intervention promoting adolescent HPV vaccination

NCT number: NCT02535845

IRB Approved date: 10-18-18

## Self-Persuasion Project Description Verbal Informed Consent Research Assistant Script (Stage 3 parent) (ENGLISH)

Thank you for agreeing to meet with me today. Before we begin, I'd like to briefly explain the study.

We are inviting parents/guardians (age 18+) of adolescents ages 9-17 with appointments at Parkland clinics to take part in this study and complete a survey. We expect about 350 people will take part.

If you agree to participate, right before your child's appointment you will use an iPad program to share your thoughts about the HPV vaccine. Then during your child's clinic appointment, we will record the conversation between doctors, nurses, and you. We will not be part of your visit, but we will leave a recorder in the room. Right after the appointment, you meet with our staff for a 20 minute recorded interview and brief survey. If your child speaks during the visit, it will be recorded. This study does not involve any medical tests or treatments. You will receive a \$50 gift card for sharing your opinions with us. In the next 12 months, the research team will look at your adolescent's medical records to see what vaccines he/she has received.

The information you provide will only be shared with members of the research team. No reports or publications by the study will use your name or other information that could identify you. There are minimal risks related to participating in this study. Some of the questions we will ask you as part of this study may make you feel uncomfortable. You may refuse to answer any of the questions, take a break or stop your participation in this study at any time. Like any research study, there is the small potential for loss of confidentiality. The information that you provide will not be reused in future research studies.

You do not have to take part in this study. If you decide to take part and later change your mind, you are free to stop at any time. Deciding <u>not</u> to take part in this study will not affect the health care you receive. By answering my questions and completing the survey, you will be consenting to participate in this study and agreeing to let the researchers have access to the information you provide.

If you have any questions about the study, please contact Dr. Jasmin Tiro's office at 214-648-0263 during regular business hours and someone will get back to you. I have a study information sheet for you which describes all of the points we've just talked about.

Do you have any questions? (Answer questions and obtain verbal informed consent and verbal HIPAA authorization from parent).

## **After parent finishes:**

Thank you for participating in this research study. In the next 12 months, the research team will look at your adolescent's medical records to see what vaccines he/she has received. If you have any further questions about the study, please contact Dr. Jasmin Tiro at number on this Study Information sheet.

**Give Study Information sheet.**